CLINICAL TRIAL: NCT05080166
Title: An Intervention for Fear of Cancer Recurrence for Lymphoma Survivors
Brief Title: UPLYFT For Lymphoma Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Society of Hematology (Other)
Responsible Party: Principal Investigator, Oreofe Odejide, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-409
Record Dates: First submitted 2021-10-05; First posted 2021-10-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma; Survivorship
Keywords: Lymphoma; Survivorship
MeSH Terms: conditions — Lymphoma | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinicians Interviews (Experimental): Lymphoma and mental health clinicians will participate in 1x in-depth qualitative interview to provide feedback for the development of the UPLYFT program.
  Interventions: Other: Interview with Clinicians
- Lymphoma Survivors Field Test (Experimental): A six person group of lymphoma survivors will participate in a six session UPLYFT program field test to provide feedback for the development of the UPLYFT program.
  Interventions: Other: Field Test of UPLYFT with Lymphoma Survivors
- UPLYFT Pilot (Experimental): Lymphoma survivors will participate in the phase 1 finalized, six session UPLYFT program.
  Participants will be randomized 1:1 to either UPLYFT or usual care.
  Interventions: Behavioral: Pilot of UPLYFT with Lymphoma Survivors

INTERVENTIONS:
Other: Interview with Clinicians — One time, qualitative interview of clinicians for feedback on UPLYFT intervention
  Arms: Clinicians Interviews
Other: Field Test of UPLYFT with Lymphoma Survivors — 6 session of UPLYFT intervention with Lymphoma Survivors for feedback
  Arms: Lymphoma Survivors Field Test
Behavioral: Pilot of UPLYFT with Lymphoma Survivors — 6 session of UPLYFT intervention with Lymphoma Survivors
  Arms: UPLYFT Pilot

SUMMARY:
The main purpose of this study is to field test and pilot an intervention called UPLYFT (Understand and Prevail: Lymphoma Fear of Recurrence Therapy) that includes information about lymphoma survivorship and tools to improve quality of life and reduce lymphoma-related worries among lymphoma survivors.

DETAILED DESCRIPTION:
This is a two phase pilot study to develop and pilot the UPLYFT (Understand and Prevail: Lymphoma Fear of Recurrence Therapy) program intervention that includes lymphoma survivorship information and acceptance and commitment therapy strategies to alleviate fear of cancer recurrence, reduce distress, and improve quality of life among lymphoma survivors.

Phase 1 will be a two-part development process of the UPLYFT program based on interview feedback from lymphoma and mental health clinicians and then feedback from a six-person group of lymphoma survivors after participation in an UPLYFT program field test. Phase 2 is a randomized pilot study using the UPLFYT program finalized in Phase 1.

Research procedures include:

* In depth interview (lymphoma and mental health clinicians)
* Screening for eligibility
* 6 weekly intervention sessions (lymphoma survivors)
* Baseline Assessments and Questionnaires (lymphoma survivors)

  74 people are expected to participate in this study with 14 in Phase 1 and 60 in Phase 2.

The American Society of Hematology is providing funding for the trial.

ELIGIBILITY:
Inclusion Criteria:

Lymphoma Survivors Phase 1 and 2:

* Diagnosis of lymphoma (indolent non-Hodgkin lymphoma, aggressive non-Hodgkin lymphoma, or classic Hodgkin lymphoma)
* Age ≥ 18 years
* Interval of 3 months to 24 months from completion of first-line treatment
* In complete remission after first line of treatment
* Clinically significant FCR (score of ≥ 16 on the validated FCR Inventory-Severity Subscale [FCRI-SS).
* Access to computer (for videoconferencing)

Lymphoma clinicians and mental health clinicians Phase 1:

* Lymphoma clinicians ≥ 1 year from oncology fellowship completion OR mental health clinicians (psychologists, social workers, psychiatrists) ≥ 1 year from completion of clinical training.
* Longitudinal clinical care for patients with lymphoma by oncologists OR provision of care for patients with cancer by mental health clinicians

Exclusion Criteria:

Lymphoma Survivors Phase 1:

* Age < 18 years
* Concurrent other malignancy
* Patients with uncontrolled/untreated psychotic disorders or untreated bipolar and borderline personality disorder (as ascertained from medical record screen).

Lymphoma Survivors Phase 2:

* Age < 18 years
* Concurrent other malignancy
* Patients with uncontrolled/untreated psychotic disorders or untreated bipolar and borderline personality disorders (as ascertained from medical record screen).

  * Our study will exclude members of the following special populations:

    * Adults unable to consent
    * Individuals who are not yet adults (infants, children, teenagers)
    * Pregnant women
    * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Enrollment Rate | Up to 6 months
  Proportion of eligible patients approached that enroll in the study.
Feasibility: Program Session Completion Rate | Up to 6 months
  Proportion of study participants randomized to the intervention arm (UPLYFT) who complete all intervention sessions.
Feasibility: Data Collection Completion Rate | Up to 6 months
  Proportion of enrolled participants who complete assigned patient-reported questionnaires during the study.

SECONDARY OUTCOMES:
Acceptability: Satisfaction Rate | Up to 6 months
  Satisfaction rate is defined as the proportion of study participants randomized to the intervention arm who are satisfied with the UPLYFT program and proportion who are likely to recommend the program.
Acceptability: Disenrollment Rate | Up to 6 months
  Disenrollment rate is defined as the proportion of eligible patients who enroll in the study who then choose to disenroll from the study.
Preliminary efficacy: Fear of Cancer Recurrence (FCR) Change | Up to 6 months
  Pre-intervention to post-intervention changes in Fear of Cancer Recurrence (FCR) measured with the Fear of Cancer Recurrence Inventory (FCRI, 42-item questionnaire), with a focus on the FCRI severity subscale.
Preliminary efficacy: Quality of Life Change | Up to 6 months
  Pre-intervention to post-intervention changes in quality of life measured with the Quality of Life- Cancer Survivor instrument (a 41-item questionnaire)
Preliminary efficacy: Anxiety Change | Up to 6 months
  Pre-intervention to post-intervention changes in anxiety as measured by the Hospital and Anxiety Scale (Anxiety subscale)
Preliminary efficacy: Depression Change | Up to 6 months
  Pre-intervention to post-intervention changes in depression as measured by the Hospital Anxiety and Depression Scale (Depression subscale)
Preliminary efficacy: Psychological inflexibility Change | Up to 6 months
  Pre-intervention to post-intervention changes in psychological inflexibility as measured by the Acceptance and Action Questionnaire-II (a 7-item scale)

CONTACTS AND LOCATIONS:
Overall Officials: Oreofe O Odejide, MD, PhD, Principal Investigator — Oreofe_Odejide@dfci.harvard.edu
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu